CLINICAL TRIAL: NCT01611610
Title: Clinical Assessment of Spinal Muscular Atrophy Type II and III
Brief Title: Clinical Assessment of Spinal Muscular Atrophy Type II and III (SMA Europe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SMA Europe
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Spinal Muscular Atrophy
Keywords: outcome measures; spinal muscular atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambulant SMA (Other)
  Interventions: Other: Functional tests
- Non-ambulant SMA (Other)
  Interventions: Other: Functional tests

INTERVENTIONS:
Other: Functional tests — The ambulant patients will perform
  * MFM (20 items)
  * Hammersmith modified module - MHMFS
  * Timed tests (time to rise from the floor,...)
  * 6 minute walk test
  * PedsQL - neuromuscular module
  Arms: Ambulant SMA
Other: Functional tests — The non-ambulant patients will perform:
  * MFM (20 items)
  * Hammersmith modified module - MHMFS
  * Upper Limb Functional Items
  * Egen Klassifikation 2 questionnaire - EK2
  * PedsQL questionnaire - neuromuscular module
  Arms: Non-ambulant SMA

SUMMARY:
The aim of this project is to establish a network of clinical teams including the major neuromuscular centers in Europe.

We plan to work together to find the best common outcome measures for the following multicenter therapeutic trials.

DETAILED DESCRIPTION:
16 patients (6 ambulant and 10 non ambulant), affected by type II and type III SMA will be enrolled and assessed at baseline and 6 and 12 months later. Non ambulant patients will be assessed using the modified version of the Hammersmith Motor Functional Scale while ambulant patients will be assessed using the extended module of the Hammersmith Motor Functional Scale and timed items, the 6 minute walk and a step activity monitor. All patients will also be assessed using the Motor Function Measure (MFM), that covers the whole range of activities for both ambulant and non ambulant patients. All measures will undergo a process of validation including inter observer reliability. This information will be most valuable for any future trial and will make the groups involved ready to participate to future collaborative studies saving a lot of time on the preliminary aspects (validation, reliability, training) that will be fulfilled by the present study. The study will also provide natural history data for a 12 month period on patients with SMA II and III.

ELIGIBILITY:
Inclusion Criteria for ambulant patients:

* age between 30 months and 24 years
* documented SMA diagnosis by genetic tests; Each should also have the determination of the SMN2 copy number
* able to walk 10 meters without support
* subject who signed an informed consent- subject affiliated to a social security system

Inclusion Criteria non ambulant patients:

* documented diagnosis of SMA by genetic tests
* not able to walk 10 meters without support
* subject affiliated to a social security system
* subject who signed an informed consent

Exclusion Criteria:

* Patient who are currently involved in other clinical trials
* severe intellectual impairment limiting the comprehension of the demanded tasks
* acute neurologic, inflammatory, infectious, endocrine, orthopedic disease in the month preceding the inclusion
* chronic neurologic (besides SMA), inflammatory, infectious, endocrine, orthopedic disease which are not a natural consequence of SMA
* spinal surgery scheduled 6 months before or within 12 months after enrollment
* pregnant women

Ages: 30 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total score of Motor Function Measure at one year | at baseline and one year after

SECONDARY OUTCOMES:
Change from baseline of Pediatric Quality of Life Inventory Score at one year | at baseline and one year after
  Pediatric Quality of Life Inventory - neuromuscular module

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Principal Investigator — Institut de Myologie